CLINICAL TRIAL: NCT00663819
Title: Efficacy of Bioabsorbable Staple Line Reinforcement in Colorectal, Coloanal and Ileoanal Anastomoses: A Prospective Randomized Study
Brief Title: Bioabsorbable Staple Line Reinforcement in Colorectal,Coloanal and Ileoanal Anastomoses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Per SAP
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-109; CS150 (Other: WL Gore)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Rectal Cancer; Ulcerative Colitis; Familial Adenomatous Polyposis; Diverticulitis
Keywords: Low anterior colon resection; Proctectomy; Proctocolectomy; Anastomosis; Rectal Cancer; Ileostomy
MeSH Terms: conditions — Rectal Neoplasms; Colitis, Ulcerative; Adenomatous Polyposis Coli; Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device (Active Comparator): GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement configured for circular staplers
  Interventions: Device: GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement
- Procedure/Surgery (Other): Procedure/Surgery: colorectal, coloanal, and ileoanal anastomotic staple line without reinforcement
  Interventions: Procedure: Staple line without reinforcement

INTERVENTIONS:
Device: GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement — Colorectal, coloanal, and ileoanal anastomotic staple line reinforcement with GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement configured for circular stapler
  Arms: Device
Procedure: Staple line without reinforcement — colorectal and coloanal anastomotic staple line without reinforcement
  Arms: Procedure/Surgery

SUMMARY:
The primary purpose of this prospective, randomized multicenter center study is to evaluate and compare the outcomes of colorectal, coloanal and ileoanal anastomoses reinforced with a bioabsorbable staple line reinforcement material compared with standard non-reinforced colorectal, coloanal and ileoanal techniques with respect to the incidence of postoperative anastomotic leakage, anastomotic stricture and time to ileostomy closure, if applicable.

DETAILED DESCRIPTION:
This is a randomized prospective trial that compares the use of GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement (CBSG) to standard stapling techniques in colorectal resections. The potential exists to utilize CBSG as a means of lowering the rate of post-operative anastomotic leakage and bleeding in high-risk colorectal, coloanal, and ileoanal anastomoses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who will undergo restorative proctectomy or proctocolectomy (<10 cm from anal verge) with a low circular stapled colorectal, coloanal or ileoanal anastomosis with or without reservoir, including treatment for rectal cancer, ulcerative colitis, familial adenomatous polyposis

  , diverticulitis, perforation of the bowel/trauma.
* Subjects undergoing Hartmann's reversal with restorative proctectomy (<10 cm from the anal verge).
* Subjects may or may not have a diverting loop ileostomy as a component of their initial surgery.
* Subjects who meet the requirements of number 1 and 2, and are being treated for rectal cancer may or may not have preoperative chemoradiation therapy in the treatment of their rectal cancer.

Exclusion Criteria:

* Subjects being treated for rectal cancer with a diagnosis of inflammatory bowel disease.
* Subjects who have significant intraoperative hypotension or cardiac events.
* Subjects with collagen vascular disease, coagulopathy, significant renal or hepatic dysfunction (creatinine >1.6 or liver enzymes > 50% upper limit of normal values).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Senagore, MD, MBA, MS, Principal Investigator — University of Southern California, Keck School of Medicine
Locations (16):
- United States (16):
  - University of South Alabama, Mobile, Alabama
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - University of South Florida-Cleveland Clinic Florida, Weston, Florida
  - Advocate Healthcare/Good Shepard Hospital, Barrington, Illinois
  - John Stroger Hospital of Cook County, Chicago, Illinois
  - Peoria Surgical Group, Peoria, Illinois
  - Colon and Rectal Surgery-NEICRS Group, Fort Wayne, Indiana
  - Kenderick Regional Center, Indianapolis, Indiana
  - Spectrum Health -Ferguson Group, Grand Rapids, Michigan
  - Duluth Clinic, Duluth, Minnesota
  - Albany Medical College, Albany, New York
  - St. Lukes-Roosevelt Hospital Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - University Hospitals of Cleveland, Case Medical Center, Cleveland, Ohio
  - Texas Endosurgery Institute, San Antonio, Texas
  - University of Utah Health Sciences Center and Huntsman Cancer Hospital, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device | Procedure/Surgery
Started | 123 | 135
Completed | 123 | 135
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients were considered for the study if they were at least 18 years of age and scheduled to undergo one the following (with the anastomosis < 10 cm from the anal verge): low anterior resection, proctectomy, proctocolectomy or a restorative anastomosis by means of Hartmann's reversal, coloanal anastomosis, or ileo-pouch-anal anastomosis.
Groups:
- GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement: GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement configured for circular staplers
  GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement: Colorectal, coloanal, and ileoanal anastomotic staple line reinforcement with GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement configured for circular stapler
- Total: Total of all reporting groups
Arm/Group | GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement | Procedure/Surgery | Total
Number analyzed (Participants) | 123 | 135 | 258
Age, Continuous [Mean (Full Range); unit: years] | 54.7 [18.8 to 83.8] | 56.1 [21.6 to 82.9] | 55.4 [18.8 to 83.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 42 | 105
  Male | 60 | 93 | 153
Region of Enrollment [Number; unit: participants]
  United States | 123 | 135 | 258

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Experience a Clinical and/or Radiologic Anastomotic Leak
Description: The primary endpoint for the study is the proportion of subjects who experience a clinical and/or radiologic anastomotic leak through 4 - 12 weeks post procedure.
Time Frame: Completion of procedure through 4-12 weeks post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Device | Procedure/Surgery
Number analyzed (Participants) | 123 | 135
Participants | 14 | 17

2. Secondary Outcome: Identify and Compare the Rate of Anastomotic Stenosis Associated With Circular Stapled Anastomoses Constructed With and Without CBSG.
Time Frame: Post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Device | Procedure/Surgery
Number analyzed (Participants) | 123 | 135
Participants | 1 | 11

3. Secondary Outcome: Determine the Rate of Significant Staple Line Hemorrhage With and Without the Use of CBSG in Circular Stapled Anastomoses
Time Frame: Post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Device | Procedure/Surgery
Number analyzed (Participants) | 123 | 135
Participants | 2 | 6

4. Secondary Outcome: Determine the Efficacy and Further Substantiate Safety of CBSG Used in Conjunction With Circular Staplers When Performing High-risk Colorectal, Coloanal, and Ileoanal Anastomoses.
Description: Compare th number of patients experiencing significant post-operative complications when performing high-risk colorectal, coloanal, and Ileoanal anastomoses across both groups studied.
Time Frame: Within 4 - 12 weeks post-surgery
Population: "Significant" Post Operative Complications
Measure: Count of Participants; unit: Participants
Arm/Group | Device | Procedure/Surgery
Number analyzed (Participants) | 123 | 135
Participants | 13 | 10

ADVERSE EVENTS:
Time Frame: Post operative Day1, Day 3, prior to hospital discharge; at 4 - 12 weeks after surgery; at 90 days post surgery
Arm/Group | GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement | Procedure/Surgery
Serious Adverse Events (participants affected / at risk) | 21/123 | 28/135
Other Adverse Events (participants affected / at risk) | 16/123 | 49/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement (N=123) | Procedure/Surgery (N=135)
Anastomotic Leak, significant (Surgical and medical procedures) | 13 (123) | 10 (135) — A total of 23 subjects developed significant anastomotic leaks
Deep organ space infection (Infections and infestations) | 3 (3) | 5 (5)
Peritonitis (Infections and infestations) | 2 (2) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 3 (3) | 12 (12)
Prolonged ileus (Gastrointestinal disorders) | 18 (18) | 22 (22)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE SEAMGUARD® Bioabsorbable Staple Line Reinforcement (N=123) | Procedure/Surgery (N=135)
Anastomotic leak, non-significant (Surgical and medical procedures) | 1 (1) | 7 (7)
Superficial wound infection (Infections and infestations) | 11 (11) | 23 (23)
Anastomotic bleeding (Surgical and medical procedures) | 2 (2) | 6 (6)
Fistula formation (General disorders) | 1 (1) | 2 (2)
Stenosis (stricture) (Surgical and medical procedures) | 1 (1) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less